CLINICAL TRIAL: NCT05607706
Title: Effect of Maternal Odor and Kangaroo Care on Serum Cortisol and Comfort Levels in Preterm Infants: a Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Alev Sivasli, assistant professor, Istanbul Nisantasi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: anka
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Preterm Birth Complication; Stress Related Disorder; Cortisol Overproduction
Keywords: preterm infant; maternal odor; kangaroo care; cortisol
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: This research; It was planned as a Randomized Controlled Experimental Study. In the study, the effect of kangaroo care and maternal odor, which are independent variables, on the toxic stress level of preterms, which is the dependent variable, was tried to be determined. The study was carried out NICU at Anka Hospital, in Gaziantep, Turkey. The sample calculation of the research was made using the "Jamovi 1.8" program. The significance level was taken as 0.05 according to the power analysis performed to determine the sufficient sample size, and it was calculated that at least 30 patients should be included in each patient group in order to have a minimum theoretical power of 0.7. The study was planned to be conducted with a total of 135 patients, with 45 patients in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): families were not allowed to enter the NICU
- Maternal Odor (Active Comparator): Babies compared only to the mother's odor
  Interventions: Behavioral: Exposure to maternal odor
- Kangaroo care (Active Comparator): Babies given kangaroo care
  Interventions: Behavioral: Exposure to maternal odor

INTERVENTIONS:
Behavioral: Exposure to maternal odor — Exposure to maternal odor; the shirt worn by the mother is put in the baby's incubator, kangaroo care; mother lays her baby naked between her breasts
  Other Names: Kangaroo care
  Arms: Kangaroo care; Maternal Odor

SUMMARY:
Aims and objectives: Studies on stress are generally aimed at young children and infants. However, in the neonatal period, "especially in preterm babies", this issue was not given enough attention and was almost completely ignored.

Background: They are exposed to different stressors. Too much stress will increase their problems in their future lives.

Design: This study was planned as a randomized study to determine the effects of Kangaroo Care and mother scent application on toxic stress in preterm infants in the Neonatal Intensive Care Unit environment and to create evidence-based recommendations regarding these applications.

Methods: Research data were collected from a total of 92 preterm babies born. Babies were divided into 3 groups, those who never met their mothers, only mother scent group and KC group. The mother's undershirt was used as the maternal odor. Vital signs, blood cortisol levels and Preterm Infant Comfort Scale scores were determined and recorded each group.The data were evaluated by statistical analysis. The CONSORT checklist for reporting qualitative research was used.

Results: In the group that never encountered mother and mother odor, Preterm Infant Comfort Scale, blood cortisol level and vital signs showed severe stress. It was found that maternal odor is effective in reducing this stress, but kangaroo care is much more effective in preventing stress.

Conclusion: if premature babies are deprived of their mother, the stress may be exposed to reaches toxic levels. It was determined that kangaroo care application during the treatment of these babies is a more effective method in reducing stress than the maternal odor application method.

Relevance to clinical practice: The results of this study will contribute to nurses' use of kangaroo care and maternal odor in the care of preterm babies to prevent stress and related complications.Therefore, it will improve the quality of care of preterm babies in the NICU.

DETAILED DESCRIPTION:
About 15 million babies are born preterm every year around the world(Blencowe et al., 2013). This corresponds to more than one in every 10 babies born alive(Lincetto & Banerjee, 2020). This situation, which is a serious problem all over the world, causes approximately 1 million children to die from complications related to preterm birth before the age of 5 years(Walani, 2020). Many of the living preterm babies also develop psychological and physical problems that require follow-up in adolescence, adulthood or lifelong (Kajantie et al., 2021; Manninen et al., 2022). Compared to term babies, preterm babies continue their lives with lower motor and neurological abilities in the later periods of their lives(Wolke et al., 2019). In addition, unlike full-term babies, hospitalization in the neonatal intensive care unit (NICU) after birth causes them to be exposed to many stress-inducing factors such as noise, nursing intervention and light (Larkin et al., 2019).

Stress is a term used to describe th eresponse of a person to both positive and negative events that he encounters daily throughout his life. Stressors can be physical, emotional, environmental or theoretical. Stressors can all affect the body's stress response equally. Stress response, also known as "fight or flight" response or general adaptation syndrome, includes physiological changes that ocur with an individual's encounter with or perceived stress. This stres response is a result of stimulation of the sympathetic nervous system resulting in a cascade of neuro-endocrine-immune responses, with reproducible physiologic effects that include an increase in respirations, heart rate, blood pressure, and overall oxygen consumption (Franke, 2014). Physiological consequences of stress, hypothalamus-pituitary-adrenal cortisol are regulated. In response to a stressor, there is an increase in the secretion of glucocorticoids, especially cortisol(Gunnar et al., 1991).There are three different types of stress. Positive stress; this type of stress is a normal part of life, a positive and normal stress response, and is essential for a child's growth and development. Positive stress responses are infrequent, short-lived, and mild. Tolerable stress; the stress that can be tolerated is more severe, frequent, or persistent. The body responds to a greater degree, and these biochemical responses have the potential to negatively affect brain architecture. Toxic stress; toxic stress leads to prolonged stimulation of the stress response with the body's inability to fully recover(Bergman, 2019a; Weber & Harrison, 2019). It differs from a normal stress response because there is a lack of caregiver support, reassurance, or emotional attachment. Inadequate caregiver support prevents the stress response from being supported or the body returning to its initial functions.This stress causes the development of many other problems in addition to the increase in the problems that will develop due to preterm birth in their future lives. Therefore, minimizing this stress is of vital importance for preterm infants and their families (WHO, 2017; Ylijoki et al., 2020).

Studies on stress are generally aimed at young children and infants. However, in the neonatal period, "especially in preterm babies", this issue was not given enough attention and was almost completely ignored. Researching this issue will help to make serious changes and corrections in the working principles of the neonatal intensive care unit. For this reason, this study was planned to determine the effects of Kangaroo Care (KC) and Maternal Odor on preterm infants on Toxic Stress and to create evidence-based recommendations about these practices in the NICU setting.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants hospitalized in the NICU for at least 15 days (babies born less than 37 weeks of gestation, greater than 28 weeks of gestation and between 1000-2500 g), babies with a first-minute Apgar score of 7 and above, and with no feeding problems, and who do not have brain-pituitary-adrenal axis problems, babies without congenital defects, and without respiratory problems (endotracheal intubation, mechanical ventilation support or nasal continuous positive airway pressure application), and with no cardiological problems, and who have not undergone surgery, and who have been given kangaroo care by a neonatal specialist, and with no suspected or no sepsis diagnosis, who are not treated with analgesics, sedatives, muscle relaxants because it may affect/pressure the stress situation, and whose mothers do not have a mental and physical problem/condition/health problem that prevents them from giving kangaroo care

Exclusion Criteria:

* constitute the research population, were determined as follows. Babies who had a health problem during the study and had a hospitalization period of less than 15 days in the NICU were excluded from the study

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Mother odor relieves stress | 6 months
  Exposing preterm infants to maternal odor reduces stress for infants in the NICU exposed to a various stressors.

SECONDARY OUTCOMES:
Kangaroo care relieves stress | 2 months
  Kangaroo care for preterm infants reduces the stress of infants in the NICU exposed to various stressors more than maternal odor

CONTACTS AND LOCATIONS:
Overall Officials: Alev Sivasli, Principal Investigator — Nisantasi University, İstanbul, Turkey
Locations (1):
- Nisantasi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: by email